CLINICAL TRIAL: NCT05848648
Title: PPK Study Based on Quantitative Pharmacology in Patients With Pamipril
Status: Recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xin Huang, Chief pharmacist, Qianfoshan Hospital
Other Study IDs: QFS-HX-2023-PMPL-001
Record Dates: First submitted 2023-04-14; First posted 2023-05-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Pamiparib
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Detect the drug concentration in the patient's blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

SUMMARY:
This is a non-intervention, prospective, one-arm, observational real-world clinical trial. The researchers plan to recruit at least 50 qualified patients. The main purpose of this study was to establish a population pharmacokinetic model of Pamiparib and to explore the correlation between its pharmacokinetic parameters and adverse reactions.

DETAILED DESCRIPTION:
In recent years, the advent of poly(ADP-ribose) polymerase(PARP) inhibitors is one of the important breakthroughs in the field of tumor-targeted therapy, and its therapeutic effect on ovarian cancer is quite significant Pamiparib is a potent, selective, oral PARP 1/2 inhibitor. In preclinical models, pamiparib demonstrated PARP-DNA complex trapping, brain penetration, antitumor activity, and inhibition of PARylation.

Therefore, at least 50 patients using pamiparib will be included. Before and after treatment, the laboratory examination data ，blood concentration ，combined medication and adverse events of the patients will be collected. The population pharmacokinetic model of pamiparib was established to evaluate the correlation between pharmacokinetic parameters and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the patient is ≥ 18 years old and less than 80 years old.
2. Receive treatment with pamipalil.
3. The patient signed a written informed consent form.

Exclusion Criteria:

1. The expected survival time may be less than the treatment cycle.
2. Is being treated with other systemic trial drugs.
3. There are other factors that the researchers think are not suitable for joining the group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients using pamipalil must sign a written informed consent before collecting blood samples.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Blood drug concentration | 6 months
  After treating with Pamipali, blood samples were collected at different time periods

SECONDARY OUTCOMES:
Correlation between blood drug concentration and adverse events | 6 months
  Try to find the relationship between pharmacokinetic parameters and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Huang Xin, Study Director — Qianfoshan Hospital
Locations (1):
- Xin Huang, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF